CLINICAL TRIAL: NCT01898819
Title: The Effect of Dexmedetomidine in Intraocular Pressure During Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2013-0195
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Steep Trendelenburg Position With Penumoperitoneum in Robot Assisted Laparoscopic Prostatectomy
Keywords: DEXMEDETOMIDINE; intraocular pressure
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): dexmedetomidine infusion from beginning of the anesthesia to just before returning to horizontal position
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator): Saline infusion from same time period.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: dexmedetomidine
Drug: saline
  Arms: saline

SUMMARY:
Intraocular pressure is significantly increase during robot-assisted laparoscopic radical prostatectomy which is performed in a steep trendelenburg position at prolonged timeds of pneumoperitoneum. Threrefore we decided to evaluate the effect of dexmedetomidine in intraocular pressure during roboti-assisted laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-II
2. obtaining written informed consent from the parents
3. aged 20-70 years who were undergoing robot- assited laparoscopic prostatectomy

Exclusion Criteria:

1. eye surgery prevoiusly
2. unstable angina or congestive heart failure
3. concomittant eye disease (glaucoma, diabetic retinophaty, cataract, retinal detachment)
4. high intraocular pressure over 30mmHg after screening test.
5. uncontrolled hypertension (diastolic bp>110mmHg)
6. bradycardia under 60bpm
7. Ventricular conduction abnormality
8. hepatic failure
9. renal failure
10. drug hyperactivity
11. neurological or psychiatric illnesses
12. mental retardation
13. patients who can't read the consent form due to illiterate or foreigner

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Influence of dexmedetomidine in intraocular pressure during robot-assisted laparoscopic prostatectomy. | change of intraocular pressure from T0 to T11 for 60mins
  T0: Pre-induciton T1: 5min after anesthesia induction T2: 5 min after establish pneumoperitoneum T3: 15min after steep trendelenburg position T4: 30min after steep trendelenburg position T5: 45min after steep trendelenburg T6: 60min after steep trendelenburg T7: 75min after steep trendelenburg T8: 5min after returning to horizontal position T9: operation end T10: 5min after tracheal extubation T11: 60min after tracheal extubation